CLINICAL TRIAL: NCT03241693
Title: Effect of a Blended-learning Programme on Physiotherapy Students´ Attitude, Knowledge and Opinions Towards Learning Professional Ethics.
Brief Title: Blended-learning in Physiotherapy: Professional Ethics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Elena Marques-Sule, Doctor in Physiotherapy, University of Valencia
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 45/FO/18/2010
Record Dates: First submitted 2017-07-25; First posted 2017-08-07 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Ethics; Attitude; Knowledge
MeSH Terms: conditions — Behavior | interventions — Ethics; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Other): Physiotherapy students
  Interventions: Other: control group
- experimental group (Experimental): Physiotherapy students
  Interventions: Other: blended-learning in ethics

INTERVENTIONS:
Other: blended-learning in ethics — Experimental group followed clinical practices in hospital centers during 8 months.
  In addition, an online specific syllabus about Professional Ethics was developed. It consisted of 6 themes and included topics as moral values, ethics and moral, bioethics and professional ethics, ecc. Six online related activities were created: to solve situations related to real clinical practices. Six face to face group sessions based on cooperative learning were planned in order to discuss ethical issues detected among clinical practices during 4 months. Students were divided in small groups, 4-5 participants each, and active participation techniques were used.
  Arms: experimental group
Other: control group — Control group followed clinical practices in hospital centers during 8 months as usual.
  In the control group, case study method was also used, thus students in control group had to create and perform a public exposition of a real clinical case about professional ethics. Cases had to be related to clinical practices in order to recognize ethical situations in the work environment. Neither online learning nor online activities were carried out.
  Arms: control group

SUMMARY:
The aim of this study was to assess the effect of a blended-learning model on physiotherapy students´ attitude, knowledge and opinions towards learning professional ethics.

A simple-blind clinical trial was performed. An eight-month blended learning program to teach professional ethics in clinical practices was worked out. An online syllabus and online activities were elaborated, whilst face to face active participation techniques were performed to discuss ethical issues detected among practices. Students´ attitudes, knowledge and opinions towards learning professional ethics were assessed. Non-parametric tests were carried out. All the participants were informed about the study and procedures, and provided written informed consent.

DETAILED DESCRIPTION:
Participants. 139 third-year degree students of Physiotherapy Degree at the University, aged between 20 and 30 years, were recruited voluntarily from September 2010 to July 2011. All enrolled participants were informed of the purpose of the study and procedures, and provided written informed consent. The study was carried out at the institution where the authors belong.

Research design. A prospective simple-blind trial was performed. After baseline assessment, participants were allocated to one of the two groups (control group, n=65; experimental group, n=64). An external assistant not involved in the study performed assignment.

Intervention. A Physiotherapy professor with over-10-year experience in Ethics and Physiotherapy performed the teaching methodology. She opened the allocation envelopes and applied the teaching methodology to the EG according to the group assignment. The intervention consisted of an eight-month blended-learning program based in professional ethics, including two phases: A) online syllabus and online activities (4 months); and B) face to face group sessions (4 months).

ELIGIBILITY:
Inclusion Criteria:

* To study the physical therapy degree at the University of Valencia

Exclusion Criteria:

* Exclusion criterion was having prior training on Ethics subject

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2011-02 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Attitude towards learning professional ethics | 8 months
  Attitude towards learning professional ethics was measured. A self-reported questionnaire of 33 items (the "Attitudes Questionnaire towards Professional Ethics in Physiotherapy", AQPEPT) was previously described by Aguilar-Rodríguez et al. A high reliability (Cronbach's alpha=0.898) was obtained. All items of the AQPEPT approached to the one-dimensionality needed in cases where attitudes are analyzed.The higher score indicated the best attitude.

SECONDARY OUTCOMES:
Knowledge towards learning professional ethics | 4 months, 8 months
  Knowledge towards learning professional ethics was assessed. A self-reported questionnaire of 19 items (the "Perceptions about Knowledge regarding Professional Ethics in Physiotherapy", PKPEP , Cronbach's alpha=0,760) was previously described by Marques-Sule et al. The higher score indicated the best knowledge.
Opinions about the blended-learning programme. | 4 months, 8 months
  Students´ opinions about the blended-learning programme were measured. Opinions about the online learning were assessed by a questionnaire comprised of eight dichotomous questions and one open question. The eight dichotomous questions aimed at evaluating if the syllabus, activities and communication system (Virtual Classroom) were considered as useful tools or not. No central options were provided to induce students to choose a positive or negative answer. Moreover, the open question aimed at adding any personal comment about the methodology. Secondly, opinions about the methodology used in the face-to-face group sessions were assessed by a questionnaire comprised of five items and one open question. Several questions about the blended-learning program were proposed: methodology of the face-to-face learning (2 items), methodology used along the study (3 items), and an open question about how to improve the teaching of professional ethics.